CLINICAL TRIAL: NCT04082494
Title: Impact on Postoperative Wellbeing in the PACU After General or Regional Anaesthesia Through Consecutive Implementation of Personalized Musical Entertainment and a Variety of Beverages. A Pre-post-post Analysis.
Brief Title: Impact on Postoperative Wellbeing in the Post-anaesthesia Care Anaesthesia (PACU) of Personalized Music and Beverages.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Stand 04.03.2019
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Complications; Postoperative Pain
Keywords: wellbeing; Postoperative Pain; postoperative disturbances after anaesthesia
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative | interventions — Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Treatment (No Intervention): No intervention is planned for the first period. "Baseline" treatment assesment.
- Music (Experimental): Optional music via internet and noise canceling headphones will be offered.
  Interventions: Device: Music via internet and noise canceling headphones
- Music and Beverages (Experimental): Additionally to the offered optional music via internet and noise canceling headphones, there will be beverages optionally offered (with and without sugar, warm or cold).
  Interventions: Device: Music via internet and noise canceling headphones; Other: Beverages

INTERVENTIONS:
Device: Music via internet and noise canceling headphones — Optional music via internet and noise canceling headphones will be offered.
  Arms: Music; Music and Beverages
Other: Beverages — Beverages will be optionally offered (with and without sugar, warm or cold).
  Arms: Music and Beverages

SUMMARY:
Postoperative disturbances for patients' well-being in the PACU after general or spinal anaesthesia will be assessed. Influence of the offer of beverages and music will be assessed regarding their wellbeing, satisfaction and pain.

ELIGIBILITY:
Inclusion Criteria:

* elective stationary adult patients capable and willing of filling out the questionnaire

Exclusion Criteria:

* participation in other studies about wellbeing influence
* incapability of filling out the questionnaire
* patients that do not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1613 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Postoperative Wellbeing | 1 day after surgery
  Assessed with the post anaesthesiological questionnaire (ANP) Wellbeing assessed with the "Anaesthesiological Questionnaire" (ANP) which is a self-rating method for the assessment of postoperative complaints and patient wellbeing. The rating scales from 0 to 3, with 0="none" and 3="strongly". Higher wellbeing values represent a better outcome.

SECONDARY OUTCOMES:
Pain assessment | approximately 2 hours after surgery
  Numeric Rating Scale (NRS) in the postanaesthesia care unit. Pain will be assessed with the (verbal) Numerical Rating Scale (NRS) and statistically evaluated for differences between the two study groups. NRS scales from 1 to 10, with 1 describing the lowest pain score and 10 the highest pain score. Lower NRS describes a better outcome.
Administered milligram of opioids for pain medication | approximately 2 hours after surgery
  Assessment of administered morphine equivalents
Postoperative complications in the postanaesthesia care unit | approximately 2 hours after surgery
  Number of participants with following complications Delirium, postoperative cognitive dysfunction, postoperative nausea and vomiting, aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Hospital LKH Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided
After publications of our data, we plan to share our data in respect of local privacy data laws.